CLINICAL TRIAL: NCT04620499
Title: A Prospective, Single-Blinded, Randomized, Multicentre Study to Evaluate the Utility, Safety, and Efficacy of Using PEER Interactive to Inform the Prescription of Medications to Subjects With a Primary Diagnosis of a Depressive Disorder
Brief Title: PEER Interactive to Inform the Prescription of Medications
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Dr. Verner Knott, Director, Clinical Neuroelectrophysiology and Cognitive Research Laboratory, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB# 2015032
Record Dates: First submitted 2016-01-29; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Electroencephalography

STUDY DESIGN:
Intervention Model Description: Group A receives treatment as usual (TAU); Group B receives access to the PEER Report (technology under investigation)
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): EEG-guided drug prescription
  Interventions: Device: EEG
- Control (No Intervention): Will receive EEG, but drugs will be prescribed as usual

INTERVENTIONS:
Device: EEG — PEER EEG
  Arms: Experimental

SUMMARY:
Improving the prescription accuracy of psychotropic medications for military personnel diagnosed with neuropsychiatric disorders is imperative to promote accelerated treatment response and recovery. This study will determine whether PEER (Psychiatric EEG Evaluation Registry) Interactive (a comparison of a quantitative electroencephalogram (QEEG) to an existing database of subject outcomes) provides an objective adjunctive tool that is more effective in guiding treatment than the current standard of practice in the treatment of military personnel suffering from non-psychotic mental illness. For this prospective, multicenter, randomized, single-blinded, controlled study, 100 participants with a primary diagnosis of a DSM-V depressive disorder, with comorbidity of non-psychotic behavioral disorders to include mild Traumatic Brain Injury (mTBI) and Post Traumatic Stress Disorder (PTSD), will be enrolled. Participants will be randomized into a control or experimental group, and all will undergo a quantitative electroencephalogram (QEEG). For the experimental group, research staff will receive an Outcome Report from PEER Interactive and will follow the guidance of the Report to inform treatment. For the control group, research staff will not receive a participant Outcome Report from PEER Interactive and these participants will be treated based on current standards. For the control group, Outcome Reports will be sequestered for post-hoc analysis. Research staff in collaboration with CNS Response (the Sponsor) will evaluate and validate if the guidance provided by PEER Interactive correlates with the predicted participant outcome. Research staff in collaboration with the Sponsor will also evaluate if the treatment guidance provided by PEER Interactive results in improved mental health and/or a reduction of risk as measured by a reduction in severe adverse events, including suicidality.

DETAILED DESCRIPTION:
Study Design

This is a prospective, single-blinded, randomized, multicenter study to evaluate the utility, safety, and efficacy of using PEER Interactive to inform the prescription of medications to participants with a primary diagnosis of a depressive disorder, with or without comorbidity of non-psychotic behavioral disorders, versus treatment as usual.

This study is observational in nature, in that the participants in the control group will be treated according to treatment as usual and best judgment of the treating clinician. The participants in the experimental group will be treated with adjunctive information provided by the PEER Interactive Report. It is a controlled study in that the schedule of visits, procedures and measurements will be defined by the protocol in order to provide consistent data for both the control and experimental groups.

Participants will be blinded as to presence/use of the PEER Interactive Report and will provide the primary efficacy outcome evaluation. All participants will be randomized into a control or experimental group. All participants will receive a quantitative electroencephalogram (QEEG). For those participants in the experimental group, the research staff will receive an Outcome Report from PEER Interactive. The clinician in the experimental group will use the PEER Interactive Report in the medication prescription process. For the control group, the research staff will not receive an Outcome Report. Outcome Reports for the control group will be sequestered for post-hoc analysis.

The research staff will incorporate the information provided by the Outcome Report from PEER Interactive in their prescription decisions. PEER Interactive provides adjunctive information to assist the treating clinician in the clinical decision process. For the experimental group the research staff is expected to follow the guidance of the subject's PEER Outcome Report as regards to the participant's responsiveness to the on-label medications noted in the Report. Although the study staff is strongly encouraged to use the guidance in the medication decision, prescription of medication is a clinical decision and will be made by the research staff. A decision to not follow the guidance of the Report should be documented and explained. In some cases, the Report may indicate sensitivity for a medication to which the subject has not been responsive in previous treatment - or - if effective for the diagnosed condition may cause/have caused an undesired side effect e.g. rash, nausea, etc. The clinician must always consider subject history in the treatment decision. We expect the Report will indicate that the participant will not be responsive to the previous treatment, and therefore, the treatment should not be prescribed. The PEER Report informs medication decisions as a part of treatment. If the only medication indicated by the report is a medication the participant has had poor experience with; the participant should be treated with another medication indicated as responsive by the Report. In the event the Report indicates the participant is not responsive to any of the on-label medications in the Report, the treating clinician may prescribe according to best clinical judgment. The research staff will note the basis for all medication decisions in the subject's treatment/study file. The only change to standard of care is the use of the PEER Report to inform medication decisions for the experimental group e.g. If a participant is receiving psychotherapy/ counseling along with medical therapy prior to enrollment, the participant will continue with all other therapies as usual.

Following the guidance of the PEER Outcome Report means prescribing any medication the report indicates the subject would be responsive to and not prescribing medications the report indicates the subject would not be responsive to. The PEER Outcome Report should be followed for up to two 'medication trials' to be considered as following the guidance of the report. A 'medication trial' is defined as prescribing a new medication to treat the subject. This includes augmentation and/or switching to a different medication. Dosing adjustments are not considered a medication trial.

The research staff, in collaboration with the sponsor, will evaluate and validate how closely the information provided by PEER Interactive correlates with post-hoc demonstrated subject medication responsiveness. The research staff, in collaboration with the sponsor will also evaluate if the information provided by PEER Interactive results in improved mental health and/or a reduction of risk as measured by a reduction in Psychiatric Specific Adverse Events, including suicidality.

Essentially, there are two evaluations being made in this study. The first is an evaluation of the clinical utility of PEER Interactive where the health outcome of participants in the experimental group (those that receive information from PEER Interactive) will be compared to the outcomes of the control group (those subjects who did not receive information from PEER Interactive). The second is a validation of the PEER Interactive outcomes database which is intended to measure post-hoc the health outcomes of participants where the research staff's pharmacotherapy decisions agreed with the output of PEER Interactive. The chart below describes these evaluations.

Focus Method Endpoints Outcome database validation Post-hoc observational Mean effect in the Agreement vs. non-Agreement group Clinical utility Prospective randomized Mean effect in Experimental vs. Control group

A QEEG is required for this study. Therefore, all participants must be washed off medications for the QEEG. Though not standard clinical practice in all settings, this is a standard requirement of the QEEG process when a QEEG study is being performed to compare participant pathophysiology to a normative database composed of non-medicated participants.

The participants will be followed for not less than 6 months after the initial treatment, or until the subject has achieved maximum medical improvement (MMI). Determination of MMI is made retrospectively e.g. we can only determine that a participant has achieved MMI following that participant's demonstration of stability on medication/in treatment as evaluated across at least two visits for example: the participant is not getting better/has stabilized and will, in the judgment of the clinician, not get better. The participant will be seen on a routine basis and assessments will be made at each interaction to evaluate the participant's improvement in mental health. The participants will be closely evaluated to determine if they are experiencing any psychiatric specific adverse events. The research staff is allowed to treat the participant according to their best medical judgment, which may include adding or changing medications, seeing the participant more frequently, or other interventions. Clinicians will be encouraged to use their best clinical judgment and best clinical practice guidelines to assess the need for transition to a new medication. All interactions and interventions will be recorded in the case report form (CRF). A second QEEG will be administered at the final/study termination visit. This second QEEG will allow for analysis to indicate treatment-related changes to the QEEG. An additional analysis will be performed to identify changes that might indicate suicidal ideation (Hunter, et al. 2010 and Iosifescu, et al. 2008). This information will be compared with findings from the participant's CHRT-SR7 questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between the ages of 18 - 65 years of age or older who speak and read English.
2. Participants able to provide written informed consent to participate in the study.
3. Participants with a primary diagnosis of a DSM-V depressive disorder, including subjects with comorbidity of a non-psychotic behavioral disorder.
4. Participants with comorbidity of mild traumatic brain injury (mTBI) are eligible for inclusion in this study. mTBI will be defined according to best clinical practice guidelines. The subject should have experienced no more than 30 minutes of loss of consciousness, less than a 24 hour alteration in consciousness or mental status, less than 24 hours of post-traumatic amnesia and a Glasgow Coma Scale (best available score in the first 24 hours) of 13 or greater.
5. Participants with comorbidity of post-traumatic stress disorder (PTSD) are eligible for inclusion in this study. A score of 45 or greater on the PTSD Checklist Military/Civilian (PCL-M/C) measurement tool will qualify a subject for inclusion of diagnosis of PTSD as a comorbid condition.
6. Able to stop non-essential medications, including drugs of abuse, for 5 half-lives of the medication(s). See Appendix B for a list of the five half-life time periods for medications.

   • The potential subject's primary care physician may be consulted to make these determinations.
7. Able to be washed out of non-essential medications within 14 days, i.e. 5 half-lives are not longer than 14 days (See Appendix B).
8. Participants will be selected from patients on the psychiatric inpatient ward, partially hospitalized patients, and psychiatric outpatients.
9. Ability to comply with the requirements of the study.

Exclusion Criteria:

1. Male and female subject less than 18 years old or greater than 65 years old
2. Participants who cannot provide written informed consent
3. Diagnosis of a psychotic disorder.
4. History of, or current, open head brain trauma.
5. Subjects with comorbidity of mild traumatic brain injury (mTBI) or traumatic brain injury (TBI) who experienced greater than 30 minutes loss of consciousness, greater than 24 hour alteration in consciousness or mental status, greater than 24 hours of post traumatic amnesia, or a Glasgow Coma Scale (best available score in first 24 hours) of less than 13.
6. Participants who, in the opinion of the research staff or medical prescriber for non-psychotropic drugs (e.g., primary care, cardiovascular, etc.), would not be good candidates to be washed out of their medications and - in the case of outpatients - are unable to washout medications and/or supplements in a period of 14 days or less.
7. Participants currently prescribed Fluoxetine when assessed for study entry (due to long metabolite half-life).
8. History of: craniotomy, cerebral metastases, cerebrovascular accident; current diagnosis of seizure disorder, schizophrenia, schizo-affective disorder, dementia, mental retardation, or major depression with psychotic features; or use of depot neuroleptics in last 12 months.
9. Clinically significant medical illness, including thyroid disorders, which cannot be remediated with medication, e.g. synthroid.
10. Participation in any other therapeutic drug study within 60 days preceding inclusion.
11. Known pregnancy and/or lactation, or intent to become pregnant during this study.
12. Chronic or acute pain requiring prescription pain medication(s) (narcotic or synthetic narcotic).
13. Candidates with any metal, shrapnel or other similar objects in the head that could affect the QEEG.
14. Candidates currently stable and considered to be at Maximum Medical Improvement (MMI) on current medications.
15. Participant has a positive urine drug screen.
16. Participant has active suicidal intent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-02; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Quick Inventory of Depressive Symptomatology-Self-Report (QIDS-SR-16) | Change from Baseline to 12 weeks to monitor change in depressive symptomatology.
  Quick Inventory of Depressive Symptomatology-Self-Report (QIDS-SR-16) is a 16-item depressive symptomatology self-report questionnaires which has been useful as a way of determining a patient's level of depression before, during, and after treatment. Questions are answered by checking off the most appropriate answer to describe how they have been feeling over the past 7 days and are scored between 0-3 points per question.
  Total score can range from 0-27 with higher values indicating worse outcomes (5 or lower: no depression, 6 to 10: mild depression, 11 to 15: moderate depression, 16 to 20: severe depression, 21 or higher: very severe depression).
  The QIDS is score as follows: Sum together the highest score out of Items 1-4, Item 5 score, highest score out of Items 6-9, sum Item 10, 11, 12, 13, and 14, highest score out of Items 15 and 16, sum all of these values for the final total score.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - The Royal, Ottawa, Ontario
  - University of Ottawa Institute of Mental Health Research, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: Yes